CLINICAL TRIAL: NCT04129853
Title: The Efficacy of the Cyberlegs Xleg During Daily Activities in People With a Unilateral Lower Limb Amputation
Brief Title: The CYBERnetic LowEr Imb coGnitive Ortho-prostheis Plus Plus, 2nd Clinical Study (CLs++)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Össur Iceland ehf (Industry); University of Ljubljana (Other); Université Catholique de Louvain (Other); Scuola Superiore Sant'Anna di Pisa (Other); Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jo Ghillebert, PhD candidate, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VUB-Brubotics
Record Dates: First submitted 2019-10-11; First posted 2019-10-17 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
Keywords: Wearable robotics; Unilateral Lower Limb Amputation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crossover (Experimental): Performing a sit to stand with the Cyberlegs Xleg and comparing with their current prosthesis.
  Interventions: Device: Cyberlegs Xleg
- Case study (Experimental): Comparing the cyberlegs xleg with other devices.
  Interventions: Device: Cyberlegs Xleg

INTERVENTIONS:
Device: Cyberlegs Xleg — Sit to stand, Stair Climbing, Slope walking, L-test, Hallway walking with the current vs. cyberlegs xleg and cyberlegs vs power knee

SUMMARY:
The aim of the project is to evaluate the efficacy of the Cyberlegs X-leg in people with a unilateral transfemoral (above the knee joint) and transtibial (under the knee joint) amputation. De Cyberlegs X-leg is in continuation of the development of the Cyberlegs gamma-prototype (B.U.N. 143201732970; FAMHP reference number: 80M0725). The Cyberlegs X-leg is a motorized prosthesis which replaces the amputated part of the leg. Our hypothesis is that people with a lower limb amputation perform daily activities (e.g. walking, stair climbing, sit to stand, et cetera) easier, more comfortable and more efficient with the X-leg compared to their current prosthesis. Assessments will be based on a holistic approach in which biomechanical, physiological and psychological parameters are determined.

DETAILED DESCRIPTION:
Study design A crossover study and a case study design.

Subjects Number of subjects 14 participants will be recruited for this study.

Inclusion criteria Age:18 - 80 year Gender: men and women Level of amputation: unilateral transfemoral or transtibial Completed the rehabilitation program Functional Medicare Classification K-level 2-4

Exclusion criteria Comorbidity (hemiplegia or neurological diseases) Stump pain or bad fit of the socket

Procedures Recruitment process Experiments will take place at the research group Human Physiology and Sports Physiotherapy of campus Etterbeek from the Vrije Universiteit Brussel (Belgium). Participants will be recruited via clinical rehabilitation centers, such as V!GO (Wetteren or Pellenberg, Belgium), Jessa hospital (Hasselt, Belgium) or via advertisement and flyers. All participants will be providing written and oral information about the experimental protocol, potential risks and benefits before giving informed consent to participate in the study.

Enrolment During a first meeting with the participant (either at home or at the laboratory) the experiment will be explained, informed consent is given, and a clinical anamnesis will occur. Eventually, appointments are made for the experiments. If necessary, a copy of the participants' current socket will be made to optimize fitting and alignment to the novel prosthesis.

Familiarization The familiarization trial aimed to accustom participants to the experimental protocol, to get used to the measurements and the novel prosthesis. Participants will get enough time (60 minutes) to perform the tests with their current and novel prosthesis and to ensure a good alignment and fitting. Participants will be fitted and aligned to the novel device by a physiotherapist and prosthetist.

Experimental protocol A (people with a transfemoral amputation) Participants with a Medicare Functional Classification K-level 2 are asked to visit the laboratory two times for a sit to stand test with their current prosthesis (first experiment) and the Cyberlegs X-leg (second experiment). During the sit to stand test (Intraclass Correlation Coefficient (ICC): 0.84-0.92), the participants will be asked to rise as often as possible from their chair in thirty seconds without support of their hands.

Experimental protocol B (people with a transfemoral and -tibial amputation) Participants with a Medicare Functional Classification K-level 3 and 4 are asked to visit the laboratory two times for four consecutive tasks with ten minutes of rest in between each task. During the stair climbing test participants' will be asked to ascend and descend a staircase. Participants start in front of the staircase and are asked to ascend and descend as fast as possible. Bilateral handrails are required to allow support when needed. The ascending phase is initiated with the prosthetic side, while the first step of the descending phase is performed with the non-involved leg. The second task is the L-test (ICC: 0.97), where participants are asked to rise from a chair, walk through an office door, turn 90 degrees, walk down a hallway, turn 180 degrees and then return in the same way to the seated position. A total distance of 20 meter will be covered. The slope walking test assesses the participants' ability to ascend and descend an inclined ramp as fast as possible. For safety reasons bilateral handrails are warranted. Participants start the test in an upright position in front of the ramp and are asked to ascend the ramp, turn around on the platform, descend the ramp and return to the starting position. Finally, a hallway six-minute walk test (ICC: 0.90 - 0.96) will be performed on a hallway at a self-selected walking speed, which closely relates to the most efficient walking speed.

These four tests will be performed in four separate case studies with the POWER knee (Össur, Reykjavik) compared to the Cyberlegs X-leg, the POWER knee compared to the Cyberlegs X-leg knee with a passive ankle joint, the current prosthesis (either passive or quasi-passive) compared to the Cyberlegs X-leg and finally a passive or quasi-passive ankle joint compared to the Cyberlegs X-leg ankle joint. In the last case study, a participant with a transtibial amputation will be included.

All appointments will take place at the same hour to counteract circadian rhythm effect, and at least 24 hours between each session will be planned to counteract mental and physical fatigue.

Outcome measures and measurement devices Physical performance determinants will be gathered in terms of duration, number of stands and normal walking speed. Biomechanical outcome measures (spatiotemporal, kinematics and kinetics) will be recorded during the different tests with a motion capture system (VICON, UK), portable singe layer sensitive walkway (GAITRite®, CIR systems, USA) and inertial measurement units (Technaid®, Spain). Outcomes from these devices include joint angels, pressure plots, cadence, step width and length, and stance and swing phases. Physiological outcome measures (cardiovascular, respiratory and electrophysiological) will be collected with a heart rate sensor (Polar® M400, H7-sensor, Finland), an ergospirometric device (K5®, Cosmed, Italy), a life monitor vest (Equivital®, USA) and electromyography device (Mini Wave®, Cometa, Italy). Outcome measures from these devices include heart rate, oxygen uptake, carbon dioxide production, ventilation, electrocardiogram, skin temperature and muscle activity (peak and mean amplitude). Psychological outcome measures like the rating of perceived exertion (score between 6-20), the visual analogue scale ( score on 100) for comfort and fatigue will be collected after the tests. The EuroQol-5D (score on 100) will be filled in before each trial. Other questionnaires will be completed during the familiarization, i.e. the mini-mental state examination (score on 30), the prosthetic evaluation questionnaire and the system usability scale.

ELIGIBILITY:
Inclusion Criteria:

* Level of amputation: unilateral transfemoral or transtibial
* Completed the rehabilitation program
* Functional Medicare Classification K-level 2-4

Exclusion Criteria:

* Comorbidity (hemiplegia or neurological diseases)
* Stump pain or bad fit of the socket

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical performance determinant | 1 year
  duration of the different tests (sec) measured with a chronometer.
Physical performance determinant | 1 year
  number of stands during the sit to stand test (number)
Physical performance determinant | 1 year
  normal walking speed (m/sec)
Biomechanical outcome measure | 1 year
  joint angels (degrees) of flexion and extension of the knee and ankle joint.
Biomechanical outcome measure | 1 year
  pressure plots of both the amputated and sound foot (N/m²)
Biomechanical outcome measure | 1 year
  cadence during the hallway walking test (steps/mine)
Biomechanical outcome measure | 1 year
  step width (cm)
Biomechanical outcome measure | 1 year
  step length (cm)
Biomechanical outcome measure | 1 year
  swing phases in % of gait cycle
Biomechanical outcome measure | 1 year
  stance phases in % of gait cycle
Electrohysiological outcome measure | 1 year
  heart rate (bpm)
Physiological outcome measure | 1 year
  oxygen uptake (ml/min)
Physiological outcome measure | 1 year
  carbon dioxide production (ml/min)
Physiological outcome measure | 1 year
  ventilation (L/min)
Electrohysiological outcome measure | 1 year
  electrocardiogram
Electrohysiological outcome measure | 1 year
  skin temperature (degees celcius)
Electrohysiological outcome measure | 1 year
  muscle activity during different movements (% of the MVC)
Psychological outcome measure | 1 year
  rating of perceived exertion (arbitrary valu between 0 and 10)
Psychological outcome measure | 1 year
  the visual analogue scale (arbitrary value between 0 (worse) and 10 (best))
Psychological outcome measure | 1 year
  the EuroQol-5D
Psychological outcome measure | 1 year
  the mini-mental state examination (arbitrary value beween 0 and 30)
Psychological outcome measure | 1 year
  the prosthetic evaluation questionnaire
Psychological outcome measure | 1 year
  the system usability scale

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No